CLINICAL TRIAL: NCT02473016
Title: A Placebo-Controlled, Single-Blind Study Evaluating the Safety and Efficacy of Nasal Carbon Dioxide for the Symptomatic Treatment of Classical Trigeminal Neuralgia
Brief Title: Nasal Carbon Dioxide for the Symptomatic Treatment of Classical Trigeminal Neuralgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capnia, Inc. (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C402
Record Dates: First submitted 2015-05-29; First posted 2015-06-16 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Trigeminal Neuralgia
Keywords: Classical Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All subjects will receive both Active (Carbon Dioxide Drug Delivery System) and Placebo. This is a single-blind study so subjects will not know the order. Subjects will receive 3 doses of active and 3 doses of placebo. One dose is a 60 second delivery of CO2 or placebo. At the discretion of the investigator, subjects may receive up to 3 additional doses of CO2.
  Interventions: Drug: Carbon Dioxide Drug Delivery System (CDDS)

INTERVENTIONS:
Drug: Carbon Dioxide Drug Delivery System (CDDS) — Doses will be administered to the nostril on the side of the trigeminal episode [ipsilateral nostril].
  Other Names: Nasal CO2; Nasal Carbon Dioxide

SUMMARY:
A placebo-controlled, single-blind study to evaluate the safety and preliminary efficacy of nasal carbon dioxide for the symptomatic treatment of classical trigeminal neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18 years of age and older.
* History of classical trigeminal neuralgia with or without persistent background facial pain, not secondary, as defined by International Classification of Headache Disorders (ICHD), third edition, beta version (ICHD-3 beta, Cephalalgia 2013).
* Diagnosis of trigeminal neuralgia (TN) for at least 60 days prior to enrollment.
* Experience pain with a score of at least 5 on a 0-10 scale during a typical TN episode as reported by subject. Note: Prior to treatment pain score must a 5 or greater on a VAS.
* History of unilateral typical TN pain predominantly in the V2 branch of the trigeminal nerve.
* Absence of a significant structural lesion (e.g., a tumor) as the cause of pain as shown in at least one neuro-imaging study.
* On stable dose of all medications, including those for the treatment of TN prevention/prophylaxis, for at least 14 days prior to baseline (including, but not limited to, verapamil, lithium, melatonin, any anticonvulsant, any systemic corticosteroid or steroid injection, occipital nerve block, other cranial or extracranial nerve block, or any neurostimulation treatment). Note: Subjects are allowed to use their usual standard of care for the acute/abortive treatment of trigeminal neuralgia attacks 60 or more minutes after the initial dose, provided it is approved by the investigator.
* Capable of completing a diary.
* Able to provide written Informed Consent.

Exclusion Criteria:

* Are unable to comply with protocol requirements.
* Have recent of alcohol or drug abuse within 2 years prior to study enrollment.
* Current major psychiatric disorder: suicidal ideation, bipolar, panic disorder, schizophrenic, or psychosis. Subjects who are documented as clinically stable and not exhibiting symptoms related to their psychiatric disorder are eligible.
* History of asthma (other than mild or intermittent).
* Have an existing serious unstable systemic disease (e.g., severe emphysema, other respiratory diseases, heart disease, etc.) that precludes participation.
* Clinically significant nasal disorder (deviated septum, presence of polyps, evidence of significant congestion, rhinitis, or other nasal abnormalities) that prevents unrestricted breathing through each nostril.
* Currently on anticoagulants or have a diagnosis of a bleeding disorder.
* Current diagnosis of fibromyalgia, temporomandibular disorders (TMD), odontogenic pain or other orofacial pain.
* Surgery for treatment of TN within 30 days prior to screening. Note: Investigator must ensure that patients who have had surgery have recovered and are not experiencing any side effects from surgery for treatment of TN
* Females who are pregnant or breast-feeding and/or plan to become pregnant or to breast-feed during study participation or within 30 days after treatment.
* Participation in a previous study with nasal CO2.
* Participation in another investigational drug study within 30 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain relief assessed on a visual analog scale (VAS) in a subject diary | Assessed through 24 hours from initial dose

SECONDARY OUTCOMES:
Percentage of subjects experiencing pain freedom at 5-60 minutes assessed on a visual analog scale (VAS) in a subject diary | Assessed through 60 minutes post intial dose
Reduction in the number of attacks (recorded in a subject diary) | Assessed through 24 hours from initial dose
Increase in duration between episodes of pain (recorded in a subject diary) | Assessed through 24 hours from initial dose
Percentage of subjects with pain relief 5-60 minutes assessed on a visual analog scale (VAS) in a subject diary | Assessed through 60 minutes post intial dose
Rescue medication usage (recorded in a subject diary) | Assessed through 24 hours from initial dose
Subject satisfaction (recorded in a subject diary) | Assessed through 24 hours from initial dose
Attack recurrence (recorded in a subject diary) | Assessed through 24 hours from initial dose
Decreased trigger sensitivity (recorded in a subject diary) | Assessed through 24 hours from initial dose
Reported Adverse Events (recorded in a subject diary and during follow up phone calls) | Up to 7 days after inital dose
Reduction in intensity of attacks (recorded in a subject diary) | Assessed through 24 hours from initial dose

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Meridien Research, Tampa, Florida
  - Columbia University Medical Center, New York, New York
  - University of Pittsbugh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - University of Virginia, Charlottesville, Virginia